CLINICAL TRIAL: NCT05302583
Title: Aromatherapy Inhaler Use for Hematopoietic Stem Cell Transplant Patient Distress
Brief Title: Aromatherapy Inhaler Use for HSCT Distress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-65140
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Cancer Distress; Cancer Coping; Hematopoetic Stem Cell Transplant; Aromatherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOC only then SOC plus Aromatherapy Inhaler (Other): 1. Participant will receive standard of care pharmacological intervention (SOC) as needed throughout the day.
  2. Participants will complete the Standard of Care Pharmacological Intervention Use Log.
  3. At between 1300 and 1500 hours, study personnel will administer the NCCN Distress Thermometer and Problem List.
  Interventions: Other: Aromatherapy Inhaler
- SOC and Aromatherapy Inhaler then SOC only (Other): 1. Participant will use the aromatherapy inhaler as needed for up to two (2) hours in the morning and complete the Aromatherapy Inhaler Use Log.
  2. At between 1300 and 1500 hours, study personnel will administer the NCCN Distress Thermometer and Problem List.
  Interventions: Other: Aromatherapy Inhaler

INTERVENTIONS:
Other: Aromatherapy Inhaler — Lavender Aromatherapy Inhaler Peppermint Aromatherapy Inhaler

SUMMARY:
The purpose of this research is to evaluate aromatherapy inhaler use and how it may impact cancer distress and coping by patients in the first few days after hematopoietic stem cell transplant (HSCT).

DETAILED DESCRIPTION:
Phase 1: Transplant Day +1, +2, or +3. Phase 2: Washout Day: Standard of care (SOC) pharmacological intervention only. Phase 3: Transplant Day +3, +4, or +5). Study Completion: Transplant Day +4, +5, or +6.

*Study activities will occur on a single day for each phase. However, a three-day window for Phases 1 and 3 will allow consideration of patients' ability to participate in the immediate post-transplant period.

ELIGIBILITY:
Inclusion Criteria:

* Autologous and Allogeneic patients admitted to E1 for planned HSCT
* Patients with hematologic malignancies requiring HSCT
* No allergies to lavender or peppermint essential oils
* Must have received chemotherapy during preparative regimen (single or multi-agent regimen)
* Adult patient over 18 years of age
* Able to speak, read, and comprehend English
* Willing and capable of providing informed consent

Exclusion Criteria:

* Patients admitted for Chimeric Antigen Receptor T cell (CART) infusion
* Patients receiving a transplant for a germ cell tumor diagnosis
* Unexpected/unplanned admission (e.g., neutropenic fever, confusion, clinical deterioration)
* Immune effector cell-associated neurotoxicity syndrome (ICANS) grade 1 through 4
* History of scleroderma
* History of atrial fibrillation
* Known history of G6PD deficiency
* Allergic to lavender or peppermint essential oils
* Pediatric patient 18 years of age or less
* Unable to speak, read, and comprehend English
* Unwilling or incapable of providing informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Attitudes and Beliefs about Complementary and Alternative Medicine Survey | Phase 1 Baseline (Transplant Day +1, +2 or +3), Phase 3 (Transplant Day +3, +4 or +5)
  15-item Likert-type scale (1 = Strongly Disagree, 5 = Strongly Agree); domain scores range between 0 and 100 and are evaluated separately; higher scores indicate greater expected benefits, perceived barriers, and positive subjective norms
Change in NCCN Distress Thermometer | Phase 1 Baseline (Transplant Day +1, +2 or +3); through Study Completion Day (Transplant Day +4, +5 or +6)
  Distress "thermometer" (visual analog scale; 0 = No Distress, 10 = Extreme Distress) for rating distress
Change in NCCN Distress Problem List | Phase 1 Baseline (Transplant Day +1, +2 or +3) through Study Completion Day (Transplant Day +4, +5 or +6)
  Distress specific problem list in five domains (checklist); optional open-ended question about "other problems"
Change in Cancer Behavior Inventory (Brief Form) | Phase 1 Baseline (Transplant Day +1, +2 or +3) through Study Completion Day (Transplant Day +4, +5, or +6)
  12-item Likert-type scale (1 = Not at all Confident, 5 = Moderately Confident, 10 = Totally Confident); rate level of confidence in range of activities, behaviors and feelings while undergoing and after cancer treatment
Aromatherapy Inhaler Use Log | Up to 6 days
  Log of aromatherapy inhaler use completed by patients.
Standard of Care Pharmacological Interventions - Nausea (STAnford Research Repository - STARR) | Up to 6 days
  Chart review using STAnford Research Repository (STARR) of pharmacological Interventions for nausea (ondansetron, lorazepam, prochlorperazine IV or oral, IV aprepitant).
Standard of Care Pharmacological Interventions - Insomnia | Phase 1 (Transplant Day +1, +2 or +3), Phase 3 (Transplant Day +3, +4 or +5)
  Chart review using STAnford Research Repository (STARR) of pharmacological Interventions for insomnia (trazodone oral, melatonin oral).
Standard of Care Pharmacological Interventions - Pain | Up to 6 days
  Chart review using STAnford Research Repository (STARR) of pharmacological Interventions for pain (oxycodone oral, hydromorphone IV or oral, IV fentanyl, acetaminophen oral, morphine IV or oral).
Final Evaluation of Aromatherapy | Study Completion Day (Transplant Day +4, +5, or +6)
  5-item Likert-type scale (1 = Terrible, 5 = Neutral, 10 = Exceptional); patient assessment of aromatherapy experience

CONTACTS AND LOCATIONS:
Overall Officials: Anna Oh, PhD, MPH, RN, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No